CLINICAL TRIAL: NCT02748746
Title: Early Detection of Lymphedema With Bio-Electrical Impedance Analysis in Patients After Breast Cancer Surgery
Acronym: BIA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to achieve device(s) which will be used in this study.
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AbantIBU
Record Dates: First submitted 2016-04-07; First posted 2016-04-22 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Lymphedema; Electric Impedance; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgery no Lymphedema (Experimental): The inclusion criteria for involving the first group is surgery time. No one will be involved into the first group if surgery was applied 18 months ago before enrollment to this study. Measurements will be done at baseline, 6th month and 12th month. Tissue dielectric constant measurement will be applied to upper extremity both affected and unaffected. 6 cm lower point of cubital crease, 8 cm upper point of cubital crease and 10 cm lower point of armpit will be marked on two sides with a soft pen before measurement. Bio impedance Analysis measurement will be done at both side. Self-adhesive electrodes will be applied related side's foot dorsum and hand dorsum. Impedance ratios will be calculated for each side then dividing process is conducted for determining L-dex ratio.
  Interventions: Device: Bio Impedance Analysis Measurement; Device: Tissue Dielectric Constant Measurement
- Surgery having Lymphedema (Experimental): The second group will contain patients who had breast cancer surgery and having upper extremity lymphedema.Measurements will be done at baseline, 6th month and 12th month. Tissue dielectric constant measurement will be applied to upper extremity both affected and unaffected. 6 cm lower point of cubital crease, 8 cm upper point of cubital crease and 10 cm lower point of armpit will be marked on two sides with a soft pen before measurement. Bio Impedance Analysis measurement will be done at both side. Self-adhesive electrodes will be applied related side's foot dorsum and hand dorsum.Impedance ratios will be calculated for each side then dividing process is conducted for determining L-dex ratio.
  Interventions: Device: Bio Impedance Analysis Measurement; Device: Tissue Dielectric Constant Measurement
- Healthy Women (Active Comparator): The third group will contain healthy women. Measurements will be done at baseline, 6th month and 12th month. Tissue dielectric constant measurement will be applied to upper extremity both affected and unaffected. 6 cm lower point of cubital crease, 8 cm upper point of cubital crease and 10 cm lower point of armpit will be marked on two sides with a soft pen before measurement. Bio Impedance Analysis measurement will be done at both side. Self-adhesive electrodes will be applied related side's foot dorsum and hand dorsum.Impedance ratios will be calculated for each side then dividing process is conducted for determining L-dex ratio.
  Interventions: Device: Bio Impedance Analysis Measurement; Device: Tissue Dielectric Constant Measurement

INTERVENTIONS:
Device: Bio Impedance Analysis Measurement — Self-adhesive electrodes will be placed to related side's hand dorsum and foot dorsum regarding to calculate for left or right upper extremity's impedance. After completing the measurements for each side, results will be saved by device and documented on paper. A patient total measurement time lasts approximately 3 minutes.
  Other Names: Bio Electrical Impedance Analysis
Device: Tissue Dielectric Constant Measurement — In this study, TDC device (Moisture Meter-D compact-MMDc will be implemented to upper extremity both affected and unaffected side. 6 cm lower point of cubital crease, 8 cm upper point of cubital crease and 10 cm lower point of armpit will be marked on two sides with a soft pen before measurement. A gentle pressure must required to have accurate sub-tissue fluid percent. Triplicate measurements will be done and taken those average value for each point in order to reach sensitive screening. Computer software simultaneously save these measurements results automatically. A patient total measurement time approximately lasts 5 minutes.
  Other Names: TDC

SUMMARY:
Bio-electrical impedance analysis and Tissue Dielectric Constant measurements are objective methods in clinical usage to detect lymphedema in early stage. The aim of this study is to reveal comparative relation these two methods on detecting lymphedema in an early stage.The another aim of this study is to determine impedance ratios and lymphedema index (L-dex) by using bio-electrical impedance analysis in patients after breast cancer surgery.

DETAILED DESCRIPTION:
Lymphedema is characterized by accumulation of protein rich fluid in interstitial spaces. It is also a chronic condition that needs lifelong care. Untreated lymphedema leads to chronic inflammation, cellulitis, pain, tiredness, cosmetic deformities, restriction of individual's motion, mobility problems and dysfunctional use of affected extremity. Undiagnosed lymphedema worsens gradually thus detecting lymphedema in an early stage have a place in matter. It was indicated that early treatment of lymphedema improves treatment outcomes.

Bio-Electrical Impedance Analysis is a non-invasive method that measures extracellular fluid proportion and impedance of related extremity by an advanced low intensity electrical current passes through body. It was stated that Bio-Electrical Impedance Analysis measures impedance ratio and it is useful in detecting lymphedema in an early stage. Bio-Electrical Impedance Analysis (BIA) gives important informations in the assessment of lymphedema by measuring directly tissue fluid changes. Lymphedema Index (L-dex) is found by dividing impedance ratios of unaffected extremity to affected extremity's impedance ratio with bio-electrical impedance analysis. Impedance of extremity lessens by developing lymphedema so L-dex value gets higher.

Tissue Dielectric Constant (TDC) is an objective and non-invasive measurement method to evaluate early tissue fluid changes. A 300 megahertz signal is generated in a control unit and transmitted to tissue by probe. Reflected electromagnetic wave depends on dielectric constant of tissue. Free and bound water molecules proportion in tissue effect tissue dielectric constant. Reflected electromagnetic wave is processed in the control unit and relative tissue dielectric constant is calculated. Dielectric constant of pure water is 78.5 in room temperature. The Scale ranges between 1-80. It was stated that comparing affected and unaffected extremities regarding lymphedema existence with TDC measurement, TDC value was higher than 1.2 in the experimental group. In the control group, TDC value was lower than 1.2 . It was also emphasized that this proportion is probably valuable on assessment of upper extremity lymphedema. TDC could be done in different depth. 0.5, 1.5, 2.5 and 5.0 mm probes are possible for usage.In this study, Moisture Meter-D compact (MMDc) device will be used for assessment. It allows evaluation in 2.5 mm depth. In this study, TDC will be applied to upper extremity both affected and unaffected side. 6 cm lower point of cubital crease, 8 cm upper point of cubital crease and 10 cm lower point of armpit will be marked on two sides with a soft pen before measurement.

Between 18-65 years old total 60 women will be recruited into the study in 3 separate groups.The first group will contain patients who had breast cancer surgery yet having no lymphedema. The inclusion criteria for involving the first group is surgery time. No one will be involved into the first group if surgery was applied 18 months ago before enrollment to this study. The second group will contain patients who had breast cancer surgery and having upper extremity lymphedema. The third group will contain healthy women. The aim of this study whether BIA and TDC methods are in capable of detecting lymphedema in an early stage. Measurements will be done at baseline, 6th month and 12th month. Exclusion criteria include being involuntary to recruit the study, bilaterally breast surgery history, having bilaterally upper extremity lymphedema, active infection, active chemotherapy and radiotherapy process, being in malignity period, and having mentally and cognitive disorders.

Lymphedema treatment may be quite costly due to materials used in the treatment and special producted compression stockings. If we take into account that compression stocking must change every six months, it carries too much importance regarding cost-effectivity that preventing lymphedema before manifesting.Even if lymphedema manifested already, detecting lymphedema in an early stage before aggravation improves treatment outcomes and individual's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being Voluntary to recruit study

Exclusion Criteria:

* Being involuntary to recruit the study
* Bilaterally Breast Surgery History
* Having Bilaterally Upper Extremity Lymphedema
* Active Infection Existence
* Active Chemotherapy
* Active Radiotherapy
* Being in Malignity Period
* Having Mentally and Cognitive Disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Investigation of early detection of lymphedema after breast cancer surgery with Bio Electrical Impedance Analysis (BIA) | 12 months
  To investigate efficacy of Bio electrical Impedance analysis method on early onset of upper extremity lymphedema.

SECONDARY OUTCOMES:
Investigation of symptom related quality of life with LymQoL | 12 months
  Symptom related quality of life questionnaire (LympQoL) will be implemented to 60 women in 3 different time frames (baseline, 6th month and 12th month). Purpose of this whether symptomatic severity changes effect the quality of life.

OTHER OUTCOMES:
Investigation of early detection of lymphedema after breast cancer surgery with Tissue Dielectric Constant (TDC) measurement | 12 months
  To investigate efficacy of Tissue Dielectric Constant (TDC) measurement method on early onset of upper extremity lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Bakar, Assoc. Prof, Study Chair — Abant Izzet Baysal University School of Physical Therapy and Rehabilitation; Alper Tuğral, Res. Assist, Principal Investigator — Abant Izzet Baysal University School of Physical Therapy and Rehabilitation; Ümmügül Üyetürk, Assoc. Prof, Principal Investigator — Abant Izzet Baysal University School of Medicine
Locations (1):
- Abant Izzet Baysal University, Bolu, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes